CLINICAL TRIAL: NCT07065604
Title: A Randomized Controlled Trial of Non-intubated Versus Intubated VATS for Mediastinal Neoplasm
Brief Title: Tubeless VATS for Mediastinal Neoplasm
Acronym: NOVA-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shuben Li (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Shuben Li, Deputy Director, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-074-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mediastinal Neoplasm; VATS; Tubeless; Non-intubated Anesthesia
Keywords: Non-intubated Anesthesia; Tubeless; Mediastinal Neoplasm; VATS
MeSH Terms: conditions — Mediastinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-intubated group (Experimental): Patients received tubeless VATS for mediastinal neoplasm
  Interventions: Procedure: Non-intubated VATS for mediastinal neoplasm
- Intubated group (Active Comparator): Patients received VATS mediastinal neoplasm resection under intubated general anesthesia.
  Interventions: Procedure: Intubated VATS for mediastinal neoplasm

INTERVENTIONS:
Procedure: Non-intubated VATS for mediastinal neoplasm — Non-intubated VATS for mediastinal neoplasm
  Arms: Non-intubated group
Procedure: Intubated VATS for mediastinal neoplasm — Intubated VATS for mediastinal neoplasm
  Arms: Intubated group

SUMMARY:
In recent year, non-intubated anesthesia had emerged as an available and promising alternative for thoracic procedure. However, its safety and feasibility in video-assisted thoracoscopic surgery (VATS) for mediastinal neoplasm remain controversial. This randomized controlled trial is designed to evaluate the impact of the non-intubated approach on surgical and perioperative outcomes in patients undergoing mediastinal neoplasm resection.

DETAILED DESCRIPTION:
Non-intubated anesthesia has gained widespread adoption in recent years, representing a significant advancement in both thoracic surgery and anesthetic practice. The surgical safety and feasibility of tubeless VATS for mediastinal neoplasm has been confirmed. However, the oncological long-term outcomes of RATS lobectomy has not been studied by randomized controlled trial. Accordingly, this randomized controlled trial aims to evaluate whether the non-intubated approach provides comparable short-term and long-term outcomes to the conventional intubated technique in VATS for mediastinal neoplasm resection.

ELIGIBILITY:
Inclusion Criteria:

1. Mediastinal neoplasm was diagnosed by chest enhanced CT
2. The patients with age ≥ 18 and ≤ 80 years old
3. The patients whose tumor diameter was <6 cm
4. ASA grade: I-III
5. The patients should understand the research and sign the informed consent

Exclusion Criteria:

1. Imaging examinations revealed that the tumor had invaded adjacent organs, with evidence of pleural or pericardial dissemination, as well as lymphatic and/or hematogenous metastases
2. Patients with a confirmed history of congestive heart failure, poorly controlled angina despite medical therapy, electrocardiogram-confirmed myocardial infarction with transmural involvement, uncontrolled hypertension, clinically significant valvular heart disease, or high-risk arrhythmias not adequately managed
3. Patients with concurrent active malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rate to open surgery | postoperative in-hospital stay up to 30 days
  Proportion of patients requiring conversion from VATS to open surgery.
Conversion rate to intubated anesthesia | postoperative in-hospital stay up to 30 days
  Proportion of patients requiring conversion from non-intubated approach to intubated anesthesia
Postoperative complication rate | postoperative in-hospital stay up to 30 days
  Incidence and severity of treatment-related adverse events, classified by Clavien-Dindo for surgical complications and CTCAE v5.0 for systemic adverse events.

SECONDARY OUTCOMES:
R0 rate | postoperative in-hospital stay up to 30 days
  R0 resection rate
Operation time | postoperative in-hospital stay up to 30 days
  Operative time was defined as the time between the start of the surgery (incision) and the finish of surgery (closure of the skin).
Intraoperative bleeding loss | postoperative in-hospital stay up to 30 days
  The volume of bleeding during the surgery.
ICU stay | postoperative in-hospital stay up to 30 days
  ICU stay (in days), defined as the duration from ICU admission post-surgery to ICU discharge.
Hospital stay | postoperative in-hospital stay up to 30 days
  Hospital stay, defined as the duration from the day of surgery to the day of discharge.
Volume of postoperative drainage | postoperative in-hospital stay up to 30 days
  Volume of postoperative drainage, measured from the end of surgery until drain removal.
1-year disease-free survival (DFS) | 1 year after surgery
  1-year disease-free survival (DFS), defined as the percentage of patients alive without evidence of tumor recurrence or progression at 12 months.
1-year overall survival(OS) | 1 year after surgery
  1-year overall survival(OS), defined as the percentage of patients alive at 12 months from the date of surgery or treatment initiation, irrespective of disease recurrence or progression.
Quality of life (QOL) at 3 month | Quality of life (QOL) at 3 months post-discharge, as measured by [specify QOL scale], reflecting patient-reported physical, emotional, and social well-being.
  3 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No